CLINICAL TRIAL: NCT06155149
Title: Effects of the Mobile Application Developed for Families Living in Tent Cities and Container Houses After the Earthquake on Burn Prevention and First Aid Knowledge and Burn Development
Brief Title: Effects of the Mobile Application Developed for Families After the Earthquake on First Aid Knowledge and Burn Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other); Harran University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Research Assistant, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TU-BOZKUL-006
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Burns; First Aid; Mobile Application; Earthquake
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm (1:1), randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A co-researcher in the project will sort the families alphabetically according to their surnames. The same co-researcher will write the number opposite each family in the list of families. An independent biostatistician, who is not involved in the study, and 30 families for each group will be determined from these numbers. Families living in container houses and tent cities were assigned to group A (control group) and group B (experimental group) by drawing lots. As a result of the draw of lots, group A will form the control group and group B will form the study group where the mobile application will be used. The data obtained from the research will be transferred to the computer environment by the other co-researcher who does not know which of the study and control groups are A and B groups. A biostatistician independent of the research will analyze the data and report the findings without knowing which of the A and B groups is the study group and which is the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): All of the families constituting the sample of the study (30 mobile application-study group) will be told about burn prevention and first aid practices with a training (powerpoint presentation) prepared by the executive researcher in line with the literature and their questions will be answered. Then, the training to be given with the mobile application will be downloaded to the phones of the families in the experimental group and the training will continue through the application.
  Interventions: Other: Mobile application; Other: Family Information Training
- CONTROL GROUP (Sham Comparator): All of the families constituting the sample of the study (30 control group) will be told about burn prevention and first aid practices with a training (powerpoint presentation) prepared by the executive researcher in line with the literature and their questions will be answered.
  Interventions: Other: Family Information Training

INTERVENTIONS:
Other: Mobile application — Mobile application: The content of the mobile application that can be used continuously after the presentation in the education of families will consist of three parts.
  In the first section: There will be short information notes and visuals on burn diagnosis and types.
  Second part: Frequently seen burns as a result of home accidents will be introduced and the precautions to be taken will be included through visuals.
  Third Section: First aid applications specific to each type of burn (scalding, fire-flame, hot contact, electrical, chemical) will be presented with visuals and information notes.
  Arms: EXPERIMENTAL GROUP
Other: Family Information Training — Family Information Training: The content of the training to be held for families in the form of a powerpoint presentation is as follows: definition of burns, classification of burns, common causes of burns at home, measures to prevent burns at home, first aid applications in burns.

SUMMARY:
The aim of this project was to determine the effect of the burn prevention and first aid mobile application developed for families living in tent cities and container houses after the earthquake on the burn prevention and first aid knowledge of families and the development of burns in the first two months after the mobile application. The research was planned as a prospective, two-arm (1:1), randomized controlled trial. The study population will consist of families living in tent cities and container houses in Şanlıurfa. As a result of the power analysis performed in the G*Power program, the sample group will consist of 30 families from the tent city and 30 families from the container city, taking into account the losses with a power of 90% and a maximum bidirectional 5% type error. All of the families (30 mobile application-study group; 30 control group) who make up the sample of the research will be given a training (powerpoint presentation) prepared by the researcher in line with the literature, and burn prevention and first aid practices will be explained and their questions will be answered. Then, the training to be given with the mobile application will be downloaded to the phones of the families in the experimental group and the training will continue through the application. In the study, data will be collected with the "Descriptive Characteristics Form", "Information Form on Burn Prevention and First Aid" and "Burn Development Follow-up Form", which include the descriptive information of the families. The data obtained from the study will be analyzed in computer environment.

DETAILED DESCRIPTION:
The aim of this project was to determine the effect of the burn prevention and first aid mobile application developed for families living in tent cities and container houses after the earthquake on the burn prevention and first aid knowledge of families and the development of burns in the first two months after the mobile application.The research was planned as a prospective, two-arm (1:1), randomized controlled trial. This randomized controlled trial will be reported according to CONSORT guidelines. The research population will consist of families living in tent cities and container houses in Şanlıurfa. As a result of the power analysis performed in the G*Power program, the sample group will consist of 30 families from the tent city and 30 families from the container city, taking into account the losses with a power of 90% and a maximum bidirectional 5% type error. All of the families (30 mobile application-study group; 30 control group) who make up the sample of the research will be given a training (powerpoint presentation) prepared by the researcher in line with the literature, and burn prevention and first aid practices will be explained and their questions will be answered. Then, the training to be given with the mobile application will be downloaded to the phones of the families in the experimental group and the training will continue through the application. Thus, families will be able to access the training from the mobile application at any time after the training. The primary results of the research are the effect of the mobile application on burn prevention and first aid knowledge. The secondary outcome of the study is the effect of the mobile application on the development of burns in the first two months after the mobile application. In the study, data will be collected with the "Descriptive Characteristics Form", "Information Form on Burn Prevention and First Aid" and "Burn Development Follow-up Form", which include the descriptive information of the families. The data obtained from the study will be analyzed in computer environment.

ELIGIBILITY:
Inclusion Criteria:

* Living in a tent-container house after the earthquake,
* No communication problems in the family,
* At least one person in the family who will participate in the training can speak Turkish,
* Written and verbal permission to participate in the study was obtained.

Exclusion Criteria:

* Not living in a tent-container house after the earthquake,
* Not wanting to participate in the research,
* The family wants to separate at any time,
* Relocation from tent cities or container houses included in the implementation area during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Burn prevention | 6 months
  Information Form on Burn Prevention and First Aid: Questions prepared by the researchers inquiring information about the training (first aid in burns, risky situations for burns, precautions to be taken, etc.).
First aid knowledge | 6 months
  Information Form on Burn Prevention and First Aid: Questions prepared by the researchers inquiring information about the training (first aid in burns, risky situations for burns, precautions to be taken, etc.).

SECONDARY OUTCOMES:
Burn development status | 2 months
  Burn Development Monitoring Form: It is a form that inquires whether burns developed within the first two months after the mobile application, and in case of development, the status of being affected by the burn and the first aid applications made.

CONTACTS AND LOCATIONS:
Overall Officials: Sabri Karahan, Study Director — Harrran University; Gülay Altun Uğraş, Principal Investigator — Mersin University; Gamze Bozkul, Principal Investigator — Tarsus University
Locations (1):
- Gamze Bozkul, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asghari Amrei S, Ayatollahi H, Salehi SH. A Smartphone Application for Burn Self-care. J Burn Care Res. 2020 Feb 19;41(2):384-389. doi: 10.1093/jbcr/irz181. PMID 31701149
- [Background] Akkoç, M. F. & Özdemir, M. (2022). Dicle Üniversitesi Yanık Merkezinde 2011-2020 Yılları Arasında Tedavi Edilen Yanık Hastalarının Epidemiyolojik Olarak İncelenmesi . Dicle Tıp Dergisi , 49 (1) , 229-235 . https://doi.org/10.5798/dicletip.1086407
- [Background] AlQahtani FA, Alanazi MA, Alanazi MK, Alshalhoub KS, Alfarhood AA, Ahmed SM. Knowledge and practices related to burn first aid among Majmaah community, Saudi Arabia. J Family Med Prim Care. 2019 Feb;8(2):594-598. doi: 10.4103/jfmpc.jfmpc_382_18. PMID 30984679
- [Background] Erkuran, M. K. , Ceylan, A. , Düzenli, E. & Büyükcam, F. (2013). Şanlıurfa Eğitim ve Araştırma Hastanesi' nde Yatırılarak İzlenmiş Olan Yanık Vakaları. Abant Tıp Dergisi, 2 (2), 123-129 . https://doi.org/10.5505/abantmedj.2013.74745 .
- [Background] Fang, T. J., Chen, H., Lee, L. C., & Wei, W. J. (2021). Development and Validation of a Mobile App for Burn Healing Care based on Interactive Design. In 2021 IEEE 4th International Conference on Knowledge Innovation and Invention (ICKII) (pp. 5-9). IEEE.
- [Background] Garcia DI, Howard HR, Cina RA, Patel S, Ruggiero K, Treiber FA, Lesher AP. Expert Outpatient Burn Care in the Home Through Mobile Health Technology. J Burn Care Res. 2018 Aug 17;39(5):680-684. doi: 10.1093/jbcr/iry013. PMID 29562343
- [Background] Güzel, A., Soyaral, L., Öncü, M., & Çakır, C. (2012). Yanık ünitemize başvuran ve cerrahi müdahale yapılan olguların incelenmesi. Van Tıp Dergisi, 19(1), 1 - 7.